CLINICAL TRIAL: NCT06622746
Title: Endoscopic Hand Suturing After Advanced Endoscopic Resections - Early Outcomes of 31 Cases in Upper and Lower GI Tract.
Brief Title: Endoscopic Hand Suturing After Advanced Endoscopic Resections.
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Zofia Orzeszko, MD, Jagiellonian University
Other Study IDs: 2024.000.586
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Endoscopic Surgical Procedures
Keywords: Endoscopic Hand Suturing; Suturing Techniques; Endoscopic Submucosal Dissection; Submucosal Tunneling Endoscopic Resection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EHS: All individuals who underwent advanced endoscopic procedures followed by EHS from March 2023 to June 2024
  Interventions: Procedure: Endoscopic Hand Suturing

INTERVENTIONS:
Procedure: Endoscopic Hand Suturing — Endoscopic Hand Suturing is a technique of the wound closure after advanced endoscopic third-space resections I the upper and lower gastrointestinal tract. In this technique, the needle is held on the opposite side from the tip with the needle holder. The needle is pierced perpendicularly into the tissue at the side of the wound with an appropriate margin, then driven through the tissue with rotation and grasped at the bottom of the defect. The same steps are repeated from the middle of the wound to create a symmetrical structure.

SUMMARY:
Endoscopic hand-suturing (EHS) has emerged as a promising modality in gastrointestinal (GI) endoscopic procedures. The available reports regarding its effectiveness in clinical practice are limited due to the relatively recent expansion of this method. This study aims to describe the single-center experience of EHS and its outcomes.

DETAILED DESCRIPTION:
Endoscopic hand-suturing (EHS) has emerged as a promising modality in gastrointestinal (GI) endoscopic procedures. The available reports regarding its effectiveness in clinical practice are limited due to the relatively recent expansion of this method. This study aims to describe the single-center experience of EHS and its outcomes. The retrospective single-center study included individuals that underwent advanced endoscopic procedures in upper and lower GI tract followed by EHS. Defined features (suturing time, suturing speed) and outcomes (postprocedural bleeding, abdominal pain) were assessed. Thirty-one patients were included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* all individuals who underwent advanced endoscopic procedures followed by EHS from March 2023 to June 2024.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective single-center study included all individuals who underwent advanced endoscopic procedures followed by EHS from March 2023 to June 2024. Procedures were conducted both in the upper and lower GI tract and included endoscopic intermuscular dissection (EID), endoscopic mucosal resection (EMR), ESD, EFTR, POEM, and STER. The EHS was performed to close a GI wall defect (after EMR, ESD, or EID) or the linear entry mucosal incision (after POEM or STER). The indications for additional suturing were high risk of bleeding following ESD in upper GI (based on patients' history of anticoagulant therapy and advanced age), closing the deep wall defect after EID in the rectum to improve recovery, closing the full-thickness defect after EFTR in cases of submucosal lesions, and concurrent treatment for perforation during ESD.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Suturing time | From 1st of March 2023 to 30th of July 2024.
  The time between delivering and retrieving the needle, in minutes.
Suturing speed | From 1st of March 2023 to 30th of July 2024.
  Calculated by dividing the longitudinal length of the defect in millimeters by the suturing time in minutes.

SECONDARY OUTCOMES:
Postprocedural bleeding rate | From 1st of March 2023 to 30th of July 2024.
  The prevalence of the symptoms of gastrointestinal bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Spychalski, PhD, Study Chair — Center of Bowel Treatment; Zofia Orzeszko, PhD, Principal Investigator — Jagiellonian University in Cracow
Locations (1):
- Jagiellonian University, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
We intend to share the encrypted data with other investigators after appropriate application and approval of the study chair.

REFERENCES:
- [Background] Goto O, Oyama T, Ono H, Takahashi A, Fujishiro M, Saito Y, Abe S, Kaise M, Iwakiri K, Yahagi N. Endoscopic hand-suturing is feasible, safe, and may reduce bleeding risk after gastric endoscopic submucosal dissection: a multicenter pilot study (with video). Gastrointest Endosc. 2020 May;91(5):1195-1202. doi: 10.1016/j.gie.2019.12.046. Epub 2020 Jan 7. PMID 31923410
- [Background] Akimoto T, Goto O, Sasaki M, Mizutani M, Tsutsumi K, Kiguchi Y, Takatori Y, Nakayama A, Kato M, Fujimoto A, Ochiai Y, Maehata T, Kaise M, Iwakiri K, Yahagi N. Endoscopic hand suturing for mucosal defect closure after gastric endoscopic submucosal dissection may reduce the risk of postoperative bleeding in patients receiving antithrombotic therapy. Dig Endosc. 2022 Jan;34(1):123-132. doi: 10.1111/den.14045. Epub 2021 Jun 22. PMID 34021512
- [Background] Uozumi T, Abe S, Mizuguchi Y, Sekiguchi M, Toyoshima N, Takamaru H, Yamada M, Kobayashi N, Sadachi R, Ito S, Takada K, Kishida Y, Imai K, Hotta K, Ono H, Saito Y. Endoscopic hand suturing using a modified through-the-scope needle holder for mucosal closure after colorectal endoscopic submucosal dissection: Prospective multicenter study (with video). Dig Endosc. 2024 Nov;36(11):1245-1252. doi: 10.1111/den.14808. Epub 2024 May 22. PMID 38775419
- [Background] Akimoto T, Goto O, Sasaki M, Mizutani M, Tsutsumi K, Kiguchi Y, Nakayama A, Kato M, Fujimoto A, Ochiai Y, Maehata T, Kaise M, Iwakiri K, Yahagi N. Endoscopic suturing promotes healing of mucosal defects after gastric endoscopic submucosal dissection: endoscopic and histologic analyses in in vivo porcine models (with video). Gastrointest Endosc. 2020 May;91(5):1172-1182. doi: 10.1016/j.gie.2019.12.032. Epub 2020 Jan 3. PMID 31904381
- [Background] Abe S, Saito Y, Tanaka Y, Ego M, Yanagisawa F, Kawashima K, Takamaru H, Sekiguchi M, Yamada M, Sakamoto T, Matsuda T, Goto O, Yahagi N. A novel endoscopic hand-suturing technique for defect closure after colorectal endoscopic submucosal dissection: a pilot study. Endoscopy. 2020 Sep;52(9):780-785. doi: 10.1055/a-1120-8533. Epub 2020 Mar 23. PMID 32207119